CLINICAL TRIAL: NCT04582162
Title: Comparison of Short Implant Assisted Mandibular Overdenture Designs (A Randomized Clinical Trial)
Brief Title: Comparison of Short Implant Assisted Mandibular Overdenture Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: short implant in overdentures
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Mandibular Bone Resorption
Keywords: short implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unsplinted implants (Experimental)
  Interventions: Other: Unsplinted implants
- Splinted implants (Active Comparator)
  Interventions: Other: Splinted implants

INTERVENTIONS:
Other: Unsplinted implants — Patients received ball abutments on each implant without splinting for retaining an implant retained mandibular overdenture.
  Arms: Unsplinted implants
Other: Splinted implants — Patients had their implants splinted using Rhein bars with ball extension for retaining an implant retained mandibular overdenture.
  Arms: Splinted implants

SUMMARY:
The aim of the study was to clinically and radiographically evaluate and compare the use of unsplinted and splinted short implants with ball abutments to support mandibular overdentures in cases with severe mandibular ridge resorption.

DETAILED DESCRIPTION:
Twelve patients from the Prosthodontics Department in the Faculty of Dentistry, Alexandria University participated in the study. Patients were divided into 2 groups. The test group received 4 short implants with ball abutments for the construction of a mandibular assisted overdenture, while the control group received 4 short implants splinted using a bar with a ball attachment for retaining a mandibular overdenture.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients.
* Mandibular ridge should be a maximum of 10mm height and with a minimum width of 8 mm to insert implants without grafting procedures.
* Patients free from systemic diseases that contradict the use of dental implants.
* Patients with class I ridge relation.
* Patients with adequate zone of keratinized mucosa.
* Patients with U-shaped or square shaped arches

Exclusion Criteria:

* Non-compliant patients based on history.
* Heavy smokers.
* Senile patients (over 75 years) with impaired neuromuscular control.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Implant stability | up to 12 months
  Stability was assessed using resonance frequency analysis measured with the Osstell device instrument. The Osstell unit records a numeric value of 1-100 which is referred to as the implant stability quotient (ISQ). The measurements were performed and 3 mean of three readings were recorded in each evaluation period.
Peri-implant probing depth | up to 12 months
  Peri-implant probing depth refers to the distance between the gingival margin and the most apically probable portion in millimeters (mm). The peri-implant probing depth was measured using a graduated plastic periodontal probe. The probe was held parallel to the long axis of the implant and introduced to the peri-implant sulcus until slight resistance was felt. Measurements were made at four sites around each implant; buccal, lingual, mesial and distal. Probing depth of 1 mm or less was recorded as "1mm", and those exceeding 1 mm but less than 2 mm were recorded as "2mm" and so forth. The mean records for each implant were then calculated.
Clinical attachment loss | up to 12 months
  It is the distance from the junction implant/abutment to the most apically probable portion, in millimeters. Assessment of the clinical attachment level was performed simultaneously while measuring the peri-implant probing depth.
Gingival inflammation (Modified gingival index) | up to 12 months
  The peri-implant mucosal tissues around the implants were assessed using Apse's modification of Löe and Silness index. The criteria for assessment were:
  0 =Normal mucosa, 1 =Mild inflammation, slight change in colour and texture, slight oedema and no bleeding on probing, 2 =Mild inflammation, redness, in all portions of gingival margin, 3 =Moderate inflammation, 4 =Severe inflammation. The gingival index was assessed at 4 sites around each implant (buccal, lingual, mesial and distal) the sum gingival index score was calculated from all these surfaces and then divided by 4 to obtain the gingival index for each implant. Indices of the three implants were added to each other, and then divided by 3 to get the mean gingival index for each case. A score from 0.1-1.0 reflects mild inflammation; 1.1-2.0 reflects moderate inflammation from, and 2.1-3.0 signifies severe inflammation.
Crestal bone loss | up to 12 months
  Mesial and Distal crestal bone loss were evaluated using digital periapical x-rays. In order to standardize the cones' and sensors' position and angulation, a film positioning system was used along with a customized silicone bite.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Weheda, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Ahmed A Abdelhakim, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Magued H Fahmy, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Nermeen A Rady, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Rocchietta I, Fontana F, Simion M. Clinical outcomes of vertical bone augmentation to enable dental implant placement: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):203-15. doi: 10.1111/j.1600-051X.2008.01271.x. PMID 18724851
- [Background] Bell RB, Blakey GH, White RP, Hillebrand DG, Molina A. Staged reconstruction of the severely atrophic mandible with autogenous bone graft and endosteal implants. J Oral Maxillofac Surg. 2002 Oct;60(10):1135-41. doi: 10.1053/joms.2002.34986. PMID 12378486
- [Background] Gentile MA, Chuang SK, Dodson TB. Survival estimates and risk factors for failure with 6 x 5.7-mm implants. Int J Oral Maxillofac Implants. 2005 Nov-Dec;20(6):930-7. PMID 16392351
- [Background] Annibali S, Cristalli MP, Dell'Aquila D, Bignozzi I, La Monaca G, Pilloni A. Short dental implants: a systematic review. J Dent Res. 2012 Jan;91(1):25-32. doi: 10.1177/0022034511425675. Epub 2011 Oct 27. PMID 22034499
- [Background] Baggi L, Cappelloni I, Di Girolamo M, Maceri F, Vairo G. The influence of implant diameter and length on stress distribution of osseointegrated implants related to crestal bone geometry: a three-dimensional finite element analysis. J Prosthet Dent. 2008 Dec;100(6):422-31. doi: 10.1016/S0022-3913(08)60259-0. PMID 19033026
- [Background] Bernard JP, Szmukler-Moncler S, Pessotto S, Vazquez L, Belser UC. The anchorage of Branemark and ITI implants of different lengths. I. An experimental study in the canine mandible. Clin Oral Implants Res. 2003 Oct;14(5):593-600. doi: 10.1034/j.1600-0501.2003.120908.x. PMID 12969363
- [Background] Stellingsma C, Meijer HJ, Raghoebar GM. Use of short endosseous implants and an overdenture in the extremely resorbed mandible: a five-year retrospective study. J Oral Maxillofac Surg. 2000 Apr;58(4):382-7; discussion 387-8. doi: 10.1016/s0278-2391(00)90917-0. PMID 10759117